CLINICAL TRIAL: NCT05733078
Title: Effect of Vitamin C Supplementation in Patients With Primary Hypothyroidism Requiring High Levothyroxine Dosage; a Randomized Control Trial
Brief Title: Effect of Vitamin C Supplementation in Patients With Primary Hypothyroidism
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr Adnan Agha (Other)
Responsible Party: Sponsor-Investigator, Dr Adnan Agha, Assistant Professor, Internal Medicine, College of Medicine and Health Sciences, United Arab Emirates University, United Arab Emirates University
Organization: United Arab Emirates University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UAEU_CMHS_IM_DOH_2023/56
Record Dates: First submitted 2023-02-02; First posted 2023-02-17 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Hypothyroidism; Primary Hypothyroidism; Vitamin C Deficiency
MeSH Terms: conditions — Hypothyroidism; Ascorbic Acid Deficiency | interventions — Ascorbic Acid

STUDY DESIGN:
Intervention Model Description: Randomization of patients:
  The patient will be randomized into control(placebo) and test (Vit C tablet) groups using the randomization code. The patients in treatment group will be provided vitamin C effervescent tablets to use 1 gram daily with their usual dose of Levothyroxine for 12 weeks. In the control group the patients will be given oral rehydration effervescent tablet as placebo with their usual dose of Levothyroxine for 12 weeks.
  The patient in test group will be provided vitamin C effervescent tablets to use 1 gram daily with their usual dose of Levothyroxine for 12 weeks, with thyroid function tests assessed at 6 and 12 weeks. The patients who wish to continue at the end of 12 weeks will be provided another 12 weeks supply of vitamin C effervescent tablets to use 1 gram daily with their usual dose of Levothyroxine for with thyroid function tests and clinical score assessed at the end of week 24.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control / Crossover (Placebo Comparator): The patients in control group will have a oral rehydration effervescent tablet to take with their usual dose of Levothyroxine for 12 weeks, with thyroid function tests assessed at 6 and 12 weeks.
  Crossover: After first 12 weeks, the control group will then be provided vitamin C (intervention) effervescent tablets to use 1 gram daily with their usual dose of Levothyroxine for 12 weeks, with thyroid function tests assessed at 6 and 12 weeks to see if there is any difference on biochemical testing or clinical scores.
  Interventions: Drug: Oral Rehydration Salt Formulations
- Intervention (Experimental): The patient in test group will be provided vitamin C effervescent tablets to use 1 gram daily with their usual dose of Levothyroxine for 12 weeks, with thyroid function tests assessed at 6 and 12 weeks. The patients who wish to continue at the end of 12 weeks will be provided another 12 weeks supply of vitamin C effervescent tablets to use 1 gram daily with their usual dose of Levothyroxine for with thyroid function tests and clinical score assessed at the end of week 24.
  Interventions: Drug: Vitamin C

INTERVENTIONS:
Drug: Vitamin C — The patient in test group will be provided vitamin C effervescent tablets to use 1 gram daily with their usual dose of Levothyroxine for 12 weeks, with thyroid function tests assessed at 6 and 12 weeks. The patients who wish to continue at the end of 12 weeks will be provided another 12 weeks supply of vitamin C effervescent tablets to use 1 gram daily with their usual dose of Levothyroxine for with thyroid function tests and clinical score assessed at the end of week 24.
  Arms: Intervention
Drug: Oral Rehydration Salt Formulations — The patients in control group will have a oral rehydration effervescent tablet to take with their usual dose of Levothyroxine for 12 weeks, with thyroid function tests assessed at 6 and 12 weeks. The control group will then be provided vitamin C (intervention) effervescent tablets to use 1 gram daily with their usual dose of Levothyroxine for 12 weeks, with thyroid function tests assessed at 6 and 12 weeks to see if there is any difference on biochemical testing or clinical scores.
  Other Names: Vitamin C
  Arms: Control / Crossover

SUMMARY:
Thyroid disease affects almost a quarter of a billion individuals worldwide and more than 50% of them being not aware of this condition. The commonest thyroid disease is iodine deficiency related thyroid dysfunction with nearly 2 billion people around the globe at risk with insufficient iodine intake. Autoimmune thyroid disorders are commonest cause of thyroid dysfunction in iodine sufficient parts of the world. Sub-optimally or untreated hypothyroidism can lead to cognitive decline, dyslipidemia, hypertension, infertility as well as cardiovascular and neuromuscular problems. The prevalence of hypothyroidism can vary in general population with up-to 5.3% people with overt hypothyroidism based on studies from the West, with estimated 10% of the population having subclinical hypothyroidism globally. In the gulf region however, there are no national studies that provide insight into exact prevalence of hypothyroidism, however some cross-sectional screening studies indicate frequency of hypothyroidism to be as high as 5-10%.

Levothyroxine is a synthetic hormone with structure similar to naturally occurring thyroxine, and it is used as replacement monotherapy of hypothyroidism. It is mainly absorbed via small intestine. The optimal daily levothyroxine dosage requirement is 1.6 microgram/kg body weight/day, which can normalize TSH in most patients, however many studies indicate that nearly half the patient on replacement therapy may not attain a normal TSH and require further doses, possibly due to interference or malabsorption. Multiple dose change and repeated diagnostic procedures in these patients can not only increased health costs but increased of ensuing complications secondary to sub-optimally controlled hypothyroidism. Instead of increasing levothyroxine doses and getting variable response, recent study have shown improvement in thyroid function by adding on vitamin C alongside levothyroxine dose, albeit only in a specific subset of patient having gastritis. The effect of Vitamin C on improving levothyroxine also been shown to be effective over a short period in a non-randomized, non-controlled setting. Our study aims to investigate whether addition of vitamin C to levothyroxine can improve the biochemical and clinical thyroid status in a randomized controlled setting.

DETAILED DESCRIPTION:
Nearly 20-50% patients with hypothyroidism do not achieve normal TSH on levothyroxine replacement and two common reasons are interference in absorption and compliance. This study aims to evaluate the effects of oral vitamin C given alongside oral levothyroxine in compliant patient with clinical/biochemical hypothyroidism despite being on optimal daily dose of levothyroxine, in terms of biochemical improvement of thyroid function status. This may help patients requiring more than recommended daily dose (> 1.6 ug/kg per day of oral levothyroxine) to achieve euthyroid status without increasing total levothyroxine dose by just adding vitamin C (which authors feel may help with improving absorption of Levothyroxine).

OBJECTIVE:

To measure the biochemical and clinical responses in thyroid status with additional oral vitamin C in patients with features of hypothyroidism who are already on recommended daily dose of >1.6 ug/kg/day of oral levothyroxine.

METHODOLOGY:

STUDY DESIGN:

This is a prospective randomized controlled study in which all adult patients known to have primary hypothyroidism, attending Tawam Hospital Endocrine clinic for the last 6 months, and fulfilling the criteria below, will be selected. We will aim to include minimum 32 patients. The study power calculations for population of Al Ain estimated 650,000 with an estimated global prevalence of hypothyroidism being around 6% and expected 20-50% (taken as 33%) with suboptimal thyroid function, indicates need for minimum 31 patient with confidence interval of 95% and margin of error as 5%. The patients will be randomized to either control or intervention group (16 in each group).

ELIGIBILITY:
Inclusion Criteria:

* Age > 18; both male or female
* Diagnosed to have Primary hypothyroidism > 6 months.
* Under follow up in Endocrine clinic in Tawam hospital during the 6 months
* No evidence of secondary hypothyroidism (no pituitary problems/surgery or thyroid surgery/ablation)
* TSH > 4 despite being on > 1.6 ug/kg/day of Levothyroxine for more than 8 weeks

Exclusion Criteria:

* Presence of coeliac disease
* Presence of selenium or iodine deficiency
* Gastric/intestinal resection surgery or confirmed malabsorption syndromes
* Known mental health issues affecting compliance
* Patient unable to consent.
* Overt biochemical hypothyroidism with TSH > 20 or T4 < 6

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Change in Thyroid function (TSH) | 24 weeks
  The primary outcome will be assessing the change in TSH levels in mIU/ml before and after supplementation the same levothyroxine dose with and without intervention (1 gram of effervescent vitamin C).
Change in Thyroid function (T4) | 24 weeks
  The primary outcome will be assessing the change in T4 levels in pmol/L before and after supplementation the same levothyroxine dose with and without intervention (1 gram of effervescent vitamin C).
Change in Thyroid function (T3) | 24 weeks
  The primary outcome will be assessing the change in T3 levels in pmol/L before and after supplementation the same levothyroxine dose with and without intervention (1 gram of effervescent vitamin C).

SECONDARY OUTCOMES:
Change in clinical status | 24 weeks
  The clinical response will be assessed by evaluating for any change in Billewicz index scoring scale questionnaires before and after intervention. Billewicz index score ≥ +25 for overt hypothyroidism; score of -30 to +25 (above -30 and below +25) for subclinical hypothyroidism; and score ≤ -30 for excluding hypothyroidism)

CONTACTS AND LOCATIONS:
Overall Officials: Adnan Agha, Principal Investigator — United Arab Emirates University
Locations (1):
- Internal Medicine, College of Medicine and Health Sciences, Al Ain City, Abu Dhabi Emirate, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Benoist B, McLean E, Andersson M, Rogers L. Iodine deficiency in 2007: global progress since 2003. Food Nutr Bull. 2008 Sep;29(3):195-202. doi: 10.1177/156482650802900305. PMID 18947032
- [Background] Jubiz W, Ramirez M. Effect of vitamin C on the absorption of levothyroxine in patients with hypothyroidism and gastritis. J Clin Endocrinol Metab. 2014 Jun;99(6):E1031-4. doi: 10.1210/jc.2013-4360. Epub 2014 Mar 6. PMID 24601693
- [Background] Virili C, Antonelli A, Santaguida MG, Benvenga S, Centanni M. Gastrointestinal Malabsorption of Thyroxine. Endocr Rev. 2019 Feb 1;40(1):118-136. doi: 10.1210/er.2018-00168. PMID 30476027
- [Derived] Agha A, Afandi B, Yasin J, Sharma C, Alshaer MH, Alshamsi MAS, Yaaqeib DE, Alblooshi BKE, AlKaabi J. Vitamin C supplementation in patients with hypothyroidism requiring high-dose levothyroxine: a proof-of-concept pilot study. Front Endocrinol (Lausanne). 2025 Oct 23;16:1679835. doi: 10.3389/fendo.2025.1679835. eCollection 2025. PMID 41210509